CLINICAL TRIAL: NCT06085261
Title: Chronic Obstructive Pulmonary Disease: A Multi-center Supervised Tele-rehabilitation Study
Brief Title: COPD: A Multi-center Supervised Tele-rehabilitation Study
Acronym: COPDMUST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ting YANG, Principal Investigator, Clinical Professor, China-Japan Friendship Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-I2M-1-409
Record Dates: First submitted 2023-08-06; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; pulmonary rehabilitation; tele-rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home-based telerehabilitation (Experimental): Remotely supervised telerehabilitation at home will be conducted for 8 weeks, comprising lower limb aerobic training, individualized strength training and respiratory training exercises.
  Interventions: Behavioral: home-based telerehabilitation group
- center-based traditional rehabilitation (Active Comparator): Participants will undertake an aerobic, strength and respiratory training program of similar intensity and duration to the home-based program, at their site of recruitment.
  Interventions: Behavioral: center-based traditional rehabilitation group

INTERVENTIONS:
Behavioral: home-based telerehabilitation group — Participants will download the web application in their smartphones in the hospital's outpatient clinic and learn to use the sports wristwatch. Remotely supervised telerehabilitation at home will be conducted for 8 weeks, comprising lower limb aerobic training, individualized strength training and respiratory training exercises. The initial aerobic exercise prescription for walking will be set at 80% of the speed walked during a 6-minute walk test (6MWT) and progressed each 4-week according to patient assessments. Resistance training for the arms and legs will utilize elastic bands, while respiratory training will utilize portable breathing trainer. During each training session, participants will be asked to follow the videos in the web application, wearing the sports wristwatch recording their exercise intensity. At the end of every training session, training data could be uploaded to the web platform automatically, which will be checked by staff in hospital.
  Arms: home-based telerehabilitation
Behavioral: center-based traditional rehabilitation group — Participants will undertake an aerobic, strength and respiratory training program of similar intensity and duration to the home-based program, at their site of recruitment.
  The initial aerobic exercise prescription for cycling will be set at 60% of the peak oxygen uptake (VO2) on a cardiopulmonary exercise test (CPET). Resistance training and respiratory training are similar to the telerehabilitation group.
  Arms: center-based traditional rehabilitation

SUMMARY:
Chronic obstructive pulmonary disease(COPD) patients could benefit from pulmonary rehabilitation(PR) in better managing of the disease and its symptoms and in avoiding future relapses and hospitalizations. However, due to a large number of drop outs from PR, lack of professionals, and the (Corona Virus Disease 2019) COVID-19 epidemic, the PR has been underutilized, leading to a need for investigation of updated forms. The study aims to investigate the effects of a home-based PR program using minimal accessories, facilitated with wearable activity trackers and smartphones.

ELIGIBILITY:
Participants with a clinical diagnosis of and meeting the following criteria are eligible:

1. Diagnosis of COPD of Global Initiative for Chronic Obstructive Lung Disease (GOLD) II-IV and without acute exacerbation within the last 2 weeks.
2. Motivated for participating in the project (and acceptance of randomization)
3. Sufficient mobility to attend PR

Exclusion Criteria:

1. Certain comorbidities (e.g. unstable coronary complications)
2. Severe cognitive disabilities (e.g. dementia)
3. Inability to cope with the program because of severe hearing or visual disorder.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) | 8 weeks; 20 weeks
  6-minute walk distance

SECONDARY OUTCOMES:
pulmonary function | 8 weeks; 20 weeks
  forced expiratory volume in 1 second (FEV1) [velocity]
pulmonary function | 8 weeks; 20 weeks
  ratio between FEV1 and forced vital capacity (FEV1/FVC) [velocity]
pulmonary function | 8 weeks; 20 weeks
  forced expiratory flow between 25 and 75% of forced vital capacity (FEF25-75%) [velocity]
pulmonary function | 8 weeks; 20 weeks
  inspiratory capacity (IC) [velocity]
pulmonary function | 8 weeks; 20 weeks
  residual volume (RV) [velocity]
pulmonary function | 8 weeks; 20 weeks
  total lung capacity (TLC) [velocity]
pulmonary function | 8 weeks; 20 weeks
  diffusing capacity of the lung for carbon monoxide (DLCO) [velocity]
Respiratory muscle strength | 8 weeks; 20 weeks
  maximum inspiratory pressure(MIP), maximum expiratory pressure(MEP)
Short Physical Performance Battery(SPPB) | 8 weeks; 20 weeks
  Test for health-related physical performance
modified British medical research council(mMRC) | 8 weeks; 20 weeks
  It is a self-reported symptom questionnaire ranging from 0-4 score, higher scores mean a worse outcome.
COPD assessment test(CAT) | 8 weeks; 20 weeks
  It is a self-reported quality of life questionnaire ranging from 0-10 score, higher scores mean a worse outcome.
St. George's Respiratory Questionnaire (SGRQ) | 8 weeks; 20 weeks
  It is a self-reported symptom questionnaire ranging from 0-100 score, higher scores mean a worse outcome.
Hospital Anxiety and Depression Scale(HADS) | 8 weeks; 20 weeks
  It is a self-reported psychological status questionnaire ranging from 0-42 score, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shiwei Qumu, Dr, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, China